CLINICAL TRIAL: NCT05697952
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of E1K After Single Dose in Patients With Knee Osteoarthritis
Brief Title: E1K Intra Articular(IA) Treatment for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ensol Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E1K-201
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E1K 1,200 ㎍/joint (Experimental): Injected 1,200 ㎍/joint/3 mL on target lesion
  Interventions: Drug: E1K 1,200 ㎍/joint
- E1K 2,400 ㎍/joint (Experimental): Injected 2,400 ㎍/joint/3 mL on target lesion
  Interventions: Drug: E1K 2,400 ㎍/joint
- Placebo (Placebo Comparator): Injected 3ml of saline on target lesion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: E1K 1,200 ㎍/joint — Injection of E1K 1,200 ㎍/joint/ml on target lesion
  Arms: E1K 1,200 ㎍/joint
Drug: E1K 2,400 ㎍/joint — Injection of E1K 2,400 ㎍/joint/ml on target lesion
  Arms: E1K 2,400 ㎍/joint
Drug: placebo — Injection of 3ml saline on target lesion
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of pain relief treatment on knee osteoarthritis when administered E1K or placebo in patients with knee osteoarthritis aged 40 to 70 to determine the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult, who is 40 years~70 years of age(inclusive of both age) at the date of consent
2. Subject who diagnosed knee osteoarthritis according to ACR criteria at screening visit, having pain in the knee and osteophyte formation in the X-ray, and one or more criteria as follows :

   * Aged >50
   * Morning stiffness < 30 minutes
   * Crepitus on knee motion
3. Prior to administration of IP, Subject with 50mm~70mm of 100mm Pain Visual Analog Scale (VAS) during activity of the knee of osteoarthritis(target lesion).
4. Subject with Grade 2 or Grade 3 on the knee osteoarthritis(target lesion) by Kellgren & Lawrence radiographic grading system
5. Subject who has pain on the knee osteoarthritis at least for 6 months before screening visit.
6. Subject who agrees not to use rescue medication within 48-hour of regular visit date.
7. Subject who agrees not to have ancillary physiotherapy
8. One-sided knee osteoarthritis subject or both-sided knee osteoarthritis subject who can designate the Target Lesion to one side, according to the follow criteria.

   * Designate the one with a higher 100 mm Pain Visual Analog Scale (VAS) than another, as the target lesion.
   * If 100 mm Pain Visual Analog Scale (VAS) is the same, designate the one with a higher Kellgren & Lawrence Grade than another, as the target lesion.
   * If both 100 mm Pain Visual Analog Scale (VAS) and Kellgren & Lawrence Grade are the same, designate the one that causes more clinical symptoms other than pain.
   * If above criteria are all the same, designate the right knee as the target lesion.
9. Subject who has voluntarily written informed consent for study participation.

Exclusion Criteria:

1. Subject who has secondary knee osteoarthritis such as inflammatory or infectious joint disease or rheumatoid arthritis.
2. Subject who has surgical history(ex. knee replacement surgery) on the knee osteoarthritis lesion(target lesion).
3. Subject who has conditions that can affect the joints(gout, recurrent caustic gout, joint fracture, primary osteochondrosis, Paget's disease, ochronosis, acromegaly, hematochromatosis, Wilson's disease, genetic disease(ex: hyperkinesia) and collagen gene related disorders.
4. Subject whose BMI greater than or equal to 30kg/m2 at screening.
5. Subject who is applicable to the followings prior to first day of IP administration.

   * Intra-articular injected hyaluronic acid, cell therapy and gene therapy within 6 months prior to IP administration
   * Intra-articular injected steroids into the knee osteoarthritis lesion(target lesion) within 3 months prior to IP administration
   * Administered NSAIDs or glucosamine, chondroitin sulfate, oral steroid within 14 days prior to IP administration.
   * Administered analgesics within 1 days prior to IP administration
6. Subject who has a psychological disorder(alcohol or drug addiction) and is judged by the investigator to have problems with the safety of the subject or to cause confusion in the interpretation of clinical trial results
7. Subject who has osteoarthritis on the other sites not knee(ex. Hip joint) or has pain due to other disorder so that the investigator determined not suitable for participation of the clinical trial.
8. Subject who has uncontrolled type 1 or type 2 diabete mellitus at screening visit(Glycated Hemoglobin (HbA1c) > 8%)
9. Subject has a positive test result for HIV antibody or hepatitis B antigen, hepatitis C antibody.
10. Subject who has malignant tumor history within 5 year prior to screening visit.
11. Subject who is participated in other clinical trials within 30 days prior to screening.
12. As a result of screening examination(laboratory or ECG, vital sign), subject who has clinically significant findings that are not suitable for participation in the clinical trials.
13. Subject who is pregnant or breastfeeding
14. Subject who does not agree to use a medically acceptable method of contraception during clinical trial.
15. Besides, in case investigator determine that subject is unsuitable for study participation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) | 12 weeks after administration of IP versus baseline
  Changes in the Sub-Scale(Pain) score of the WOMAC questionnaire

SECONDARY OUTCOMES:
Pain VAS 100mm | at 4, 8, and 12 weeks after administration of IP versus baseline
  Changes in 100 mm Pain VAS (Pain during activity and at rest during the last 24 hours) scores
WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) | at 4, 8, and 12 weeks after IP administration compared to baseline
  Changes in scores by WOMAC questionnaire total score and Sub-Scale (physical function, stiffness)
WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) | at 4 to 8 weeks after administration of IP compared to the baseline
  Changes in the Sub-Scale(Pain) score of the WOMAC questionnaire
KOOS | at 4, 8, and 12 weeks after administration of IP compared to baseline
  Changes in KOOS questionnaire scores
Quality of life(EQ-5D-5L) | at 4, 8, and 12 weeks after administration of IP compared to baseline
  Changes in EQ-5D-5L questionnaire scores
Frequency of Rescue drug | Day 0 to Day 84
  Percentage and number of subjects who took the rescue medication during the clinical trial period

CONTACTS AND LOCATIONS:
Overall Officials: Young-Wan Moon, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No